CLINICAL TRIAL: NCT02449200
Title: A Randomised Controlled Trial of Multimodal Physiotherapy for Patients With Acute / Sub-acute Cervical Radiculopathy
Brief Title: RCT of Multimodal Physiotherapy for Acute / Sub-acute Cervical Radiculopathy
Acronym: PACeR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal College of Surgeons, Ireland (Other)
Collaborators: Beaumont Hospital (Other); EuroSpine - the Spine Society of Europe (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GR 14-0917
Record Dates: First submitted 2015-05-05; First posted 2015-05-20 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2018-05

CONDITIONS: Cervical Radiculopathy
Keywords: cervical radiculopathy; exercise; manual therapy; tape
MeSH Terms: conditions — Radiculopathy; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multimodal physiotherapy group (Experimental): 4 week multimodal physiotherapy treatment programme provided by an experienced musculoskeletal physiotherapist
  Interventions: Other: Multimodal physiotherapy
- Advice to stay active group (No Intervention): Advice to stay active and continue use of prescribed medication as appropriate, via weekly phone calls from a physiotherapist over a 4 week period.

INTERVENTIONS:
Other: Multimodal physiotherapy — Manual therapy, exercise and neural unloading tape provided twice weekly over 4 weeks by an experienced musculoskeletal physiotherapist
  Arms: Multimodal physiotherapy group

SUMMARY:
Multimodal physiotherapy involving manual therapy and exercise has demonstrated a positive effect on pain and disability in sub-acute and chronic cervical radiculopathy (CR) but a research gap exists for optimal management in the first 12 weeks and short-term natural history of the condition is unclear, although thought to be favourable within the first 4 weeks. The primary aim of this single blind, 2 group randomised controlled trial (RCT) is to investigate the effects of a 4 week (6-8 sessions) programme of manual therapy, exercise and upper limb unloading tape compared to advice to stay active, on disability, pain and other biopsychosocial measures, in acute / sub-acute cervical radiculopathy patients. The hypothesis is that a 4 week multimodal physiotherapy programme will lead to changes in self-reported disability and pain, compared to advice to stay active, in patients with acute / sub-acute cervical radiculopathy. A secondary study objective is to identify whether variables from the baseline examination, group allocation and aetiology confirmed by MRI can predict outcome, as measured with the Global Rating of Change Scale (GROC). Subjects will be diagnosed with CR based on a diagnostic clinical prediction rule. Random group allocation, allocation concealment, blinded assessment and intention to treat analysis will be employed. Outcomes will be measured at baseline, 4 and 12 weeks. Patients' report of pain, disability and their rating of recovery will also be recorded by telephone interview at 6 months. An internal pilot feasibility study will be undertaken in advance of the main study to test recruitment and retention strategies. Statistical analysis of differences between groups will be done with ANOVAs and MANOVAs. Appropriate multivariable regression analysis will be used to explore predictors of outcome.

DETAILED DESCRIPTION:
Cervical radiculopathy (CR) has been defined by the North American Spine Society (NASS) as pain in a radicular pattern in one or both upper extremities related to compression and/or irritation of one or more cervical nerve roots, with signs and symptoms including varying degrees of sensory, motor, and reflex changes in addition to dysaesthesia and paraesthesia (Bono et al. 2011). CR is of particular clinical concern, given the higher levels of pain and disability associated with the presence of nerve-related arm pain resulting in higher healthcare costs for this cohort of people with neck pain (Rubinstein et al., 2007, Haldeman et al., 2008).

Multimodal physiotherapy involving manual therapy and exercise has demonstrated a positive effect on pain and disability for chronic (symptom duration > 3 months) CR (Boyles et al., 2011). No consensus on the optimum conservative management, or indeed optimal timing of such management, currently exists for acute / sub-acute cervical radiculopathy. The combined use of manual therapy with exercise for this cohort is now garnering interest; evident by the emergence of several randomised controlled trials (Nee et al., 2012, Langevin et al., 2015) involving treatment duration of 2-4 weeks. Langevin et al. (2015) demonstrated that using 2 varied programmes of manual therapy & exercise, led to similarly clinically significant improvements in pain and disability, particularly immediately after a 4 week intervention. However, without a 'no treatment' control group, natural recovery could not be excluded, confirming the need for adequate control groups in future trials (Langevin et al., 2015). The most recent Cochrane review of exercise for the treatment of mechanical neck disorders (MND) (including CR) concluded that there was low quality evidence to suggest a small pain reduction benefit with cervical stretch / strengthening / stabilization exercises in the short term in acute cervical radiculopathy (Gross et al., 2015). They also advocated for larger sample sizes and longer follow-up periods in future trials.

A randomised controlled trial of a 4 week course of a multimodal physiotherapy package (manual therapy (to spinal joints), exercise (mobility exercise, deep neck flexor and scapular muscle training), upper limb unloading tape (to offload the brachial plexus) and advice to stay active) for acute/sub-acute CR is proposed. As there is no strong evidence establishing best clinical practice for the conservative management of acute/sub-acute CR, a control group of advice to stay active and medication will be used.

Aims & Objectives:

The primary aim of this trial is to investigate the effects of a 4 week multimodal physiotherapy (MP) programme on neck and arm pain and resulting disability in CR, over 6 months, with the primary endpoint at 4 weeks.

Secondary objectives are:

* to investigate the effects of the MP programme on the following additional biopsychosocial outcome measures;

  * Cervical range of motion
  * Upper Limb Neurodynamic Test (ULNT) 1
  * Pressure Pain Thresholds (PPT)
  * Quality of Life
  * Anxiety and Depression
  * Fear Avoidance beliefs
  * Patient rating of recovery
* to identify whether any of the above biopsychosocial outcome measures, as well as the PainDETECT at baseline, symptom duration and group allocation; can predict outcome at 3 months, on the GROC scale.

Hypothesis:

A 4 week multimodal physiotherapy programme will lead to changes in self-reported disability and pain, compared to advice to stay active, for acute / sub-acute cervical radiculopathy.

Research Design:

An exploratory, assessor-blinded, randomised controlled trial is planned.

Procedure:

A consecutive sample of all new (non-urgent) patients with cervical radiculopathy referred by their general practitioner for neurosurgical assessment to Beaumont Hospital are being recruited.

Eligibility assessment includes a neurological exam and manual exam of the cervical spine (C2-T2) to identify the nerve root level and to guide the treating physiotherapists for those participants subsequently assigned to the intervention group. If eligible and upon providing written consent, prior to baseline assessment and random group allocation, each participant will be asked by the PI about their beliefs regarding the likely effectiveness of physiotherapy, as well as their belief in the need for surgery. Participants will be randomly assigned to the intervention or control group by an independent academic colleague using a computer-generated list of random numbers with a random block size of 4, 6 or 8.

Participants allocated to the control group will be advised to continue taking their prescribed or over the counter medication, as well as to stay active, by the treating physiotherapist. They will be telephoned weekly for 4 weeks.

Participants allocated to the intervention group will attend the Physiotherapy Department of Beaumont Hospital or Collins Avenue Physiotherapy clinic for a 4 week programme of multi-modal physiotherapy involving advice, manual therapy, exercise and upper limb unloading tape, as decided by the treating physiotherapist from a best-practice physiotherapy treatment guide. Participants in the intervention group will be treated twice a week for 30 minutes each session and receive non-provocative manual therapy (all participants will receive lateral glide mobilisation (Vicenzino et al., 1999) to the mechanical interface of the radiculopathy and additional Maitland joint mobilisation to the segmental levels above or below (as far as T4) as deemed necessary by the treating physiotherapist based on their mobility assessment), exercise (all participants will receive deep neck flexor strengthening and scapular orientation exercise as deemed necessary by the treating physiotherapist based on their motor control assessment (Jull et al., 2008)) and cervical mobility exercises. Upper limb neural unloading tape will be applied at the end of the treatment session. The tape will run from the upper arm, over the top of the shoulder and across to the back of the neck and will unload the brachial plexus. Experienced senior physiotherapists with a master's degree in musculoskeletal physiotherapy (or equivalent) will provide the treatment programme. Treating physiotherapists will also record the participants' adherence with a home exercise programme by administering a weekly exercise adherence questionnaire to monitor the participant's home exercise frequency per week.

Medication usage of participants in both groups will be monitored on a weekly basis.

In the case of a significant adverse event (progressive neurological signs e.g. multilevel or bilateral radiculopathy, myotomal paresis < 4/5 on MRC scale; or emerging medical red flags or cervical spondylotic myelopathy) during the trial, an appropriate clinical pathway will be followed. The clinical change will be discussed with the neurosurgical registrar and requirement for a fast track clinical review will be determined. Minor adverse events will also be recorded during the trial.

Participants from both groups will be assessed by the principal investigator at the end of treatment at 4 weeks and again at 12 weeks. Participants' report of pain and disability and their rating of recovery will also be recorded by telephone interview at 6 months. Baseline demographics will be recorded including co-morbidities, educational level, smoking status, occupation and work status and any change in to work status at subsequent assessment time points will be noted.

Participants will be asked not to pursue other treatment during the trial, until after the 12 week assessment. All other interventions received will be recorded at the 6 months telephone follow up.

Sample size estimation:

The NDI and the NPRS are the co-primary outcome measures for this study and sample size estimates were carried out for both outcome measures. An MCID for the NDI of 7 has been determined for cervical radiculopathy patients (Cleland et al., 2006). Using a reported NDI SD of 9.2 (Cleland et al., 2006) for this patient group, with a two-sided 5% significance level and a power of 80%, a sample size of 29 participants per group will be necessary. An MCID for the NPRS of 2 has been determined for mechanical neck pain, including cervical radiculopathy (Cleland et al., 2008) and a SD of 1.85 (Cleland et al., 2006). Using these figures, with a two-sided 5% significance level and a power of 80%, a sample size of 15 per group was calculated. The larger sample size per group calculated using the NDI was chosen and an additional 10% was added to account for anticipated dropout. In total, a sample size of 64 participants will be recruited.

Pilot study:

A pilot feasibility study will be undertaken, with the objectives of testing the recruitment strategy and retention rates of the study. The pilot study will mirror the protocol of the main study except the assessment time points will be limited to baseline and 4 weeks (at the end of treatment for the intervention group) and the pilot will run for 2 months or until the first 6 participants have reached their 4 week assessment.

Criteria for assessing success of this feasibility study (Thabane et al., 2010) will be:

* 6 participants can be recruited per month. To recruit the sample size estimate over a 12 month period, more than 5 participants per month will need to be recruited.
* Complete follow-up is possible in at least 95% of all recruited participants.

The pilot study will also identify if a difference in retention rates exists between groups, by following participants until the 4 week assessment point. Participants in the control group will also be asked how acceptable they would find continuing with medication and advice to stay active for a further 8 weeks, to assess the likelihood of dropout before the second and third assessment time points. Results from the pilot study will be included in the main study results if no further significant protocol changes are required after the pilot.

A second recruitment pathway, via direct general practitioner (GP) referral from primary care commenced during the pilot in October 2015, as it was clear the initial recruitment strategy was inadequate. This pathway was approved by the Irish College of General Practitioners Research Ethics Committee in September 2015. Five physiotherapy treatment sites are now providing the intervention across the greater Dublin area. An additional private physiotherapy practice site was added in January 2016 and 3 further physiotherapy practice sites were added in September 2016, in order to roll out the trial across Dublin.

Data analysis:

Baseline demographic characteristics and all outcome measures will be described and presented for both groups following the CONSORT Statement. Data will be checked for normality using the Shapiro-Wilk test. Marginal effects will be used to calculate effect sizes for specified values for baseline differences between the 2 groups. Poisson regression will be used where data are non-parametric.

Statistical analysis will include two-way (treatment x time) ANOVAs and MANOVAs for between and within-group differences and interactions. Intention to treat analysis will be the primary approach employed. A secondary per protocol analysis will also be undertaken.

Secondary analysis to explore if any of the outcome measures or group allocation are predictors of outcome (GROC score at 3 months) will be performed using appropriate multivariable regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for CR diagnosis on a clinical prediction rule (CPR) by demonstrating positive responses to at least 3 of the following 4 clinical tests: Spurling's Test, Upper Limb Neural Tissue Provocation Test 1 (ULNT 1), Cervical Distraction Test, and less than 60° of cervical rotation on the symptomatic side (Wainner et al., 2003).
* Complaints of neck / periscapular pain, in addition to radicular pain, paraesthesia or numbness in the upper limb; aggravated by neck posture or movement (Thoomes et al., 2012).
* Symptom duration must be greater than 2 weeks and less than 3 months.
* Mean of Numerical Pain Rating Scale (NPRS) scores for both neck and arm pain must be ≥ 3/10.
* Fluent in spoken and written English.
* Willing to give informed consent.

Exclusion Criteria:

* Previous physiotherapy / manual treatment to cervical spine within past 6 months.
* Previous epidural injection since the onset of current symptoms.
* Prior surgery to the cervicothoracic spine or currently symptomatic upper limb.
* Current symptoms & signs of bilateral radiculopathy.
* Myotomal paresis less than 4 / 5 on Medical Research Council Scale in affected upper limb.
* Signs and symptoms suggestive of Cervical Spondylotic Myelopathy (CSM): bilateral paraesthesia, hyperreflexia, positive Babinski reflex and spasticity.
* Diagnosis of any generalised neurological disorder e.g. multiple sclerosis.
* Concurrent peripheral neuropathy affecting either upper limb e.g. carpal tunnel syndrome, thoracic outlet syndrome.
* Medical red flags suggestive of serious pathology such as neoplastic conditions, upper cervical ligamentous instability, vertebral artery insufficiency and inflammatory or systemic disease (Childs et al., 2004).
* Diagnosis of fibromyalgia.
* Psychiatric diagnosis in past 6 months.
* Ongoing litigation relating to cervical symptoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2015-05 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in neck and arm pain (Numerical Pain Rating Scale) | 4 weeks
  Neck and arm pain levels measured with the Numerical Pain Rating Scale for current, best and worst pain levels over last 24 hours (Jensen et al 1994)
Change from baseline in Neck Disability Index | 4 weeks
  Disability resulting from the cervical radiculopathy measured with the Neck Disability Index (Vernon and Mior 1991)

SECONDARY OUTCOMES:
Cervical range of motion (ROM) measured with a CROM 3 device | Baseline, 4 weeks and 12 weeks
  Cervical ROM measured with a CROM 3 device (Performance Attainment Associates, USA). Flexion, extension, bilateral sideflexion and rotation will be measured.
SF-12 version 2 Health Survey | Baseline, 4 weeks and 12 weeks
  Quality of Life using the SF-12 version 2 Health Survey (Cheak-Zamora et al, 2009)
Pressure Pain Thresholds measured with a SenseBox pressure algometer | Baseline, 4 weeks and 12 weeks
  Pressure pain thresholds measured with a SenseBox pressure algometer (Somedic, Sweden) at standardised sites on both hands at site of maximal pain and anterior tibia as a remote site (Walton et al 2011).
Hospital Anxiety Depression Scale | Baseline, 4 weeks and 12 weeks
  Hospital Anxiety Depression Scale (HADS), a validated scale that assesses non-somatic symptoms of anxiety and depression (Zigmond and Snaith, 1983).
Upper Limb Neurodynamic test 1 | Baseline, 4 weeks and 12 weeks
  Upper limb neurodynamic test 1 is a validated pain provocation test of nervous tissue directly assesses nerve mechanosensitivity (Elvey, 1994 and Wainner and Gill, 2000). It is considered positive if it reproduces arm pain with differentiation tests. Degrees of elbow flexion at point of symptom onset, measured with a universal goniometer.
Fear Avoidance Belief Questionnaire (Neck) | Baseline, 4 weeks and 12 weeks
  Fear Avoidance Belief Questionnaire (FABQ). The FABQ was initially established to measure how patients' beliefs about physical activity and work affected their low back pain (Waddell et al., 1993). Landers et al. (2008) have since established that the FABQ can predict neck pain patients who may develop prolonged disability.
painDETECT Questionnaire | Baseline
  PainDETECT is a self-report questionnaire that was designed to detect neuropathic pain components in adult patients with low back pain (Freynhagen et al., 2006). It has since been used in a cervical radiculopathy cohort and will be used in this study in the secondary analysis of predictors to treatment response.
Change from baseline in neck and arm pain levels (Numerical Pain Rating Scale) | 12 weeks and 6 months
  NPRS described above
Change from baseline in Neck Disability Index | 12 weeks and 6 months
  NDI described above

CONTACTS AND LOCATIONS:
Overall Officials: Louise Keating, MPhtySt, Principal Investigator — Royal College of Surgeons in Ireland
Locations (1):
- Beaumont Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bono CM, Ghiselli G, Gilbert TJ, Kreiner DS, Reitman C, Summers JT, Baisden JL, Easa J, Fernand R, Lamer T, Matz PG, Mazanec DJ, Resnick DK, Shaffer WO, Sharma AK, Timmons RB, Toton JF; North American Spine Society. An evidence-based clinical guideline for the diagnosis and treatment of cervical radiculopathy from degenerative disorders. Spine J. 2011 Jan;11(1):64-72. doi: 10.1016/j.spinee.2010.10.023. PMID 21168100
- [Background] Boyles R, Toy P, Mellon J Jr, Hayes M, Hammer B. Effectiveness of manual physical therapy in the treatment of cervical radiculopathy: a systematic review. J Man Manip Ther. 2011 Aug;19(3):135-42. doi: 10.1179/2042618611Y.0000000011. PMID 22851876
- [Background] Childs JD, Cleland JA, Elliott JM, Teyhen DS, Wainner RS, Whitman JM, Sopky BJ, Godges JJ, Flynn TW; American Physical Therapy Association. Neck pain: Clinical practice guidelines linked to the International Classification of Functioning, Disability, and Health from the Orthopedic Section of the American Physical Therapy Association. J Orthop Sports Phys Ther. 2008 Sep;38(9):A1-A34. doi: 10.2519/jospt.2008.0303. Epub 2008 Sep 1. PMID 18758050
- [Background] Cleland JA, Childs JD, Whitman JM. Psychometric properties of the Neck Disability Index and Numeric Pain Rating Scale in patients with mechanical neck pain. Arch Phys Med Rehabil. 2008 Jan;89(1):69-74. doi: 10.1016/j.apmr.2007.08.126. PMID 18164333
- [Background] Cleland JA, Fritz JM, Whitman JM, Palmer JA. The reliability and construct validity of the Neck Disability Index and patient specific functional scale in patients with cervical radiculopathy. Spine (Phila Pa 1976). 2006 Mar 1;31(5):598-602. doi: 10.1097/01.brs.0000201241.90914.22. PMID 16508559
- [Background] Gross A, Kay TM, Paquin JP, Blanchette S, Lalonde P, Christie T, Dupont G, Graham N, Burnie SJ, Gelley G, Goldsmith CH, Forget M, Hoving JL, Bronfort G, Santaguida PL; Cervical Overview Group. Exercises for mechanical neck disorders. Cochrane Database Syst Rev. 2015 Jan 28;1(1):CD004250. doi: 10.1002/14651858.CD004250.pub5. PMID 25629215
- [Background] Haldeman S, Carroll L, Cassidy JD, Schubert J, Nygren A; Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. The Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders: executive summary. Spine (Phila Pa 1976). 2008 Feb 15;33(4 Suppl):S5-7. doi: 10.1097/BRS.0b013e3181643f40. No abstract available. PMID 18204400
- [Background] Jull, G., Sterling, M., Falla, D., Treleaven, J. & O'Leary, S. 2008. Whiplash, Headache and Neck Pain. Research-based directions for physical therapists., Churchill Livingstone.
- [Background] Langevin P, Desmeules F, Lamothe M, Robitaille S, Roy JS. Comparison of 2 manual therapy and exercise protocols for cervical radiculopathy: a randomized clinical trial evaluating short-term effects. J Orthop Sports Phys Ther. 2015 Jan;45(1):4-17. doi: 10.2519/jospt.2015.5211. PMID 25420010
- [Background] Nee RJ, Vicenzino B, Jull GA, Cleland JA, Coppieters MW. Neural tissue management provides immediate clinically relevant benefits without harmful effects for patients with nerve-related neck and arm pain: a randomised trial. J Physiother. 2012;58(1):23-31. doi: 10.1016/S1836-9553(12)70069-3. PMID 22341379
- [Background] Rubinstein SM, Pool JJ, van Tulder MW, Riphagen II, de Vet HC. A systematic review of the diagnostic accuracy of provocative tests of the neck for diagnosing cervical radiculopathy. Eur Spine J. 2007 Mar;16(3):307-19. doi: 10.1007/s00586-006-0225-6. Epub 2006 Sep 30. PMID 17013656
- [Background] Thabane L, Ma J, Chu R, Cheng J, Ismaila A, Rios LP, Robson R, Thabane M, Giangregorio L, Goldsmith CH. A tutorial on pilot studies: the what, why and how. BMC Med Res Methodol. 2010 Jan 6;10:1. doi: 10.1186/1471-2288-10-1. PMID 20053272
- [Background] Vicenzino B, Neal R, Collins D, Wright A. The displacement, velocity and frequency profile of the frontal plane motion produced by the cervical lateral glide treatment technique. Clin Biomech (Bristol). 1999 Oct;14(8):515-21. doi: 10.1016/s0268-0033(99)00011-x. PMID 10521635
- [Derived] Keating L, Treanor C, Sugrue J, Meldrum D, Bolger C, Doody C. A randomised controlled trial of multimodal physiotherapy versus advice for recent onset, painful cervical radiculopathy - the PACeR trial protocol. BMC Musculoskelet Disord. 2019 Jun 1;20(1):265. doi: 10.1186/s12891-019-2639-4. PMID 31153362
- See also: PACeR trial website — http://www.rcsi.ie/PACeRtrial